CLINICAL TRIAL: NCT00405379
Title: A Prospective Randomized Controlled Trial Using Roentgen Stereophotogrammetric Analysis of Trabecular Metal Mesh Tibial Monoblock Knee Arthroplasty Component "TMM".
Brief Title: Trabecular Metal Mesh Tibial Monoblock RSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Stryker Trauma and Extremities (Industry)
Responsible Party: Dr. Michael Dunbar MD, FRCSC, PhD, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAL06-02; CDHA-RS/2002-096
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Osteoarthritis
Keywords: arthroplasty; RSA; Osteoarthritis; trabecular metal mesh
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Trabecular Metal Mesh Tibial Monoblock Knee Arthroplasty — new porous metal tibial component with potential to result in improved bone in-growth and implant integration with proximal tibia

SUMMARY:
Trabecular Metal(TM) is a relatively new technology and its use in knee replacement is quite different from the more conventional total knee replacement (arthroplastie). The aim of incorporating TMM into the material used for the knee replacement (tibial prostheses) is to improve initial fixation of the prosthesis at the time of implantation (surgery) and to improve long term prosthesis survival by encouraging and improving bone ingrowth.

DETAILED DESCRIPTION:
Hip and knee replacement arthroplasty are profoundly successful operative interventions, however, some joint replacements do fail and the life expectancy of a hip or knee arthroplasty is finite (Malchau et al. 1993, Knutson et al. 1994, Herberts et al. 1997, Garellick et al. 1998). This fact has largely been responsible for the continued development of new devices and techniques for joint arthroplasty surgery. Unfortunately, the introduction of new technologies and devices is not a benign process, and even subtle changes to existing implants can have a disastrous effect on patient outcome (Sudmann et al. 1983, Herberts P. 1986, Ohlin et al. 1989, Wedderkopp et al. 1997, Howie et al. 1998, Nilsson et al. 1998).

The fact that new technologies and devices can lead to poor results has led some authors to advocate a phased introduction of new technologies (Gross 1988, Gross 1993, Malchau 1999). A key component of the phased introduction approach advocates the use of roentgen stereophotogrammetric analysis (RSA) early in the testing process (Malchau 1999).

RSA is a highly accurate radiographic technique developed in Lund, Sweden and has for some time been the gold standard in Europe for assessing the stability of implants within bone (Selvik 1990, Ryd 1992, Catani et al. 1998, Alfaro-Adrian et al. 1999). It is at least ten times more accurate than conventional radiography (Ryd et al. 1986). RSA involves the insertion of small tantalum markers (0.8mm) into the bone and prosthesis at the time of surgery (Ryd 1986, Ryd et al. 1986, Ryd et al. 1989, Selvik 1990, Ryd 1992). By using a calibrated cage with additional markers and simultaneous bi-planar x-rays, micromotion at the prosthesis-bone interface can be very precisely determined (Selvik et al. 1983). Two types of micromotion can be investigated: migration, i.e. gradual motion over time, and inducible displacement, i.e. instant motion in response to external forces (Ryd et al. 1986). The pattern of micromotion exhibited by various prostheses and fixation techniques within the first post-operative year has been shown to be predictive of the long-term fixation of the component to bone, especially when considering the tibial prosthesis-bone interface (Ryd 1986, Ryd et al. 1986, Ryd 1992, Ryd et al. 1995). The value of this precise radiographic technique is that new technologies and techniques can be introduced in vivo while limiting their exposure to as few patients as possible. RSA is a proven, safe and invaluable method for assessing methods of tibial component fixation as well as different design concepts (Ryd et al. 1987, Nilsson et al. 1991, Ryd et al. 1992, Ryd et al. 1993, Hilding et al. 1995, Onsten et al. 1998, Nilsson et al. 1999).

Until recently, RSA technology has been cumbersome and expensive. However, significant advances have made the system more applicable due to the fact that digitized films are being used, and computer programs have been written and can run on small personal computers that will allow for automatic capture and interpretation of x-ray markers and implants (Vrooman et al. 1998).

Trabecular Metal(TM) is a relatively new technology and its use in tibial knee arthroplasty components represents a significant departure from conventional total knee arthroplasties. TM has a high co-efficient of friction and high affinity for bone ingrowth (Bobyn et al. 1999a, Bobyn et al. 1999b, Hacking et al. 2000), subsequently, the aims of incorporating TMM into tibial prostheses is to improve initial fixation of the tibial prosthesis at the time of implantation and to improve long term prosthesis survival by facilitating bone ingrowth. Such advantages remain, however, theoretical, and have yet to be demonstrated in vivo for total knee arthroplasty. With conventional study techniques, a definitive answer to the effect of the prosthetic design on fixation of the tibial component would require a large number of patients and approximately 10 years of follow-up (Ryd 1992, Ryd et al. 1995). RSA provides a means of accurately assessing the tibial component fixation, both immediate and long term, on a relatively small number of patients within two years of the onset of the study. It is critical at this stage to determine the long-term effect of this design concept on component fixation so that any deleterious effects can be addressed and any advantageous effects can be disseminated to the orthopaedic community.

ELIGIBILITY:
Inclusion Criteria:

* Age between 55 and 80
* Primary osteoarthritis of the knee
* Mono-articular disease (Charnley Modified Type A)

Exclusion Criteria:

* Significant co-morbidity affecting ability to ambulate
* Flexion contracture greater than 15°
* Tibial subluxation greater than 10 mm on standing AP radiograph
* Greater than 10° of varus or 15° of valgus
* Extension lag greater than 10°
* Lateral or medial collateral ligament instability (> 10° varus/valgus)
* Previous osteotomy about the knee
* Previous arthroplasty of the knee
* Previous patellectomy
* Posterior cruciate ligament deficiency
* Leg length discrepancy greater than 10 mm
* Morbid obesity

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2002-07; Primary Completion 2006-08 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
micromotion of tibial component | 2 years postoperative

SECONDARY OUTCOMES:
subjective outcomes measured with health outcome questionnaires sf36, WOMAC | 2 years postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Dunbar, MD FRCSC PhD, Principal Investigator — Dalhousie University & Capital Districk Health Authority

REFERENCES:
- [Derived] Astephen Wilson JL, Wilson DA, Dunbar MJ, Deluzio KJ. Preoperative gait patterns and BMI are associated with tibial component migration. Acta Orthop. 2010 Aug;81(4):478-86. doi: 10.3109/17453674.2010.501741. PMID 20809746